CLINICAL TRIAL: NCT00321477
Title: NK1 Receptor Antagonist vs Placebo in the Treatment of Overactive Bladder Symptoms
Brief Title: A Study Of GW679769 Compared To Placebo In Women With Overactive Bladder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NKB105022
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Incontinence, Urinary and Urinary Bladder, Overactive; Overactive Bladder
Keywords: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — casopitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW679769 oral tablets

SUMMARY:
This is a Phase IIa study to evaluate the efficacy, safety and tolerability of GW679769 vs placebo on symptoms of urgency with urge incontinence, frequency and nocturia associated with overactive bladder in women.

DETAILED DESCRIPTION:
A Twelve-Week Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Forced Titration, Proof of Concept Study to Assess the Efficacy, Safety and Tolerability as well as the Pharmacokinetic Profile of 60 mg and 120 mg of GW679769 administered once daily vs Placebo in Women with Overactive Bladder

ELIGIBILITY:
Inclusion Criteria:

* Female subjects with overactive bladder with symptoms of urgency with urge incontinence and frequency which may be associated with nocturia but without bladder pain.
* Must not be pregnant.
* Must not be of childbearing potential or is willing to use specific barrier methods outlined in the protocol.
* Body weight in the range of = 45 kg and <100 kg.

Exclusion Criteria:

* Stage III/IV pelvic organ prolapse with or without cystocele.
* History of interstitial cystitis or bladder related pain.
* Subjects with stress incontinence or mixed incontinence where stress incontinence is the predominant component based on prior history.
* History of pelvic prolapse repair (cystocele or rectocele) or urethral diverticulectomy within six months of screening.
* Subjects with urinary incontinence due to causes other then detrusor over activity (e.g., overflow incontinence).
* Nocturnal enuresis only.
* Urinary retention, or other evidence of poor detrusor function.
* History of prior anti-incontinence surgery.
* History of radiation cystitis or a history of pelvic irradiation.
* Electrostimulation, biofeedback, or bladder training therapy (behavioral therapy) during the previous month prior to screening, or the intention to initiate such therapies during the study. Pessaries and implants are also excluded.
* Participated in any clinical trial of an investigation drug that may affect urinary function within 3 months of enrollment into the study.
* Received any investigational product within 30 days of enrollment into the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2005-12; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline to Week 12 in the number of incontinence episodes/24 hrs | 12 weeks

SECONDARY OUTCOMES:
Change from baseline to Weeks 6 and 12 in the following endpoints: Number of micturitions/24 hrs Number of urgency episodes/24 hrs Number of nocturia episodes/24 hrs | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (55):
- United States (39):
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Peoria, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, La Mesa, California
  - GSK Investigational Site, Modesto, California
  - GSK Investigational Site, San Bernardino, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Longmont, Colorado
  - GSK Investigational Site, Waterbury, Connecticut
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Melrose Park, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Jeffersonville, Indiana
  - GSK Investigational Site, Newburgh, Indiana
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Kingston, New York
  - GSK Investigational Site, Poughkeepsie, New York
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Springfield, Oregon
  - GSK Investigational Site, Bala-Cynwyd, Pennsylvania
  - GSK Investigational Site, Lancaster, Pennsylvania
  - GSK Investigational Site, Sellersville, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Tacoma, Washington
- Canada (16):
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Fredericton, New Brunswick
  - GSK Investigational Site, Saint John, New Brunswick
  - GSK Investigational Site, Kentville, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Barrie, Ontario
  - GSK Investigational Site, Kitchener, Ontario
  - GSK Investigational Site, Newmarket, Ontario
  - GSK Investigational Site, North Bay, Ontario
  - GSK Investigational Site, Oakville, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Pointe-Claire, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec